CLINICAL TRIAL: NCT06421389
Title: Precise Endoscopic Application of Tranexamic Acid and Sucralfate in Gastrointestinal Bleeding: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Hsueh-Chien Chiang, Attending physician, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-BR-113-014
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2024-07

CONDITIONS: Bleed Ulcer
Keywords: Bleeding ulcer; Sulcralfate; Tranexamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): All patients will receive the standard endoscopic hemostasis by either epinephrine injection, hemoclipping, heat coagulation, or band ligation. After then, patients in intervention group will receive 2g of sucralfate powder, 1g of tranexamic acid powder, and 1g of barium spray through the endoscopy precisely on the bleeding site.
  Interventions: Drug: Tranexamic Acid Powder
- Control group (No Intervention): All patients will receive the standard endoscopic hemostasis by either epinephrine injection, hemoclipping, heat coagulation, or band ligation.

INTERVENTIONS:
Drug: Tranexamic Acid Powder — 2g of sucralfate powder, 1g of tranexamic acid powder, and 1g of barium will be sprayed through the endoscopy precisely on the bleeding site
  Other Names: sucralfate powder; barrium sulfate powder
  Arms: Intervention group

SUMMARY:
Background and Aim: Gastrointestinal bleeding (GIB) is a common problem in the hospital. GIB can be divided into upper GIB, small bowel bleeding, and lower GIB. Endoscopic hemostasis includes epinephrine injection, hemoclipping, heat probe coagulation, and Argon plasma coagulation. Although the successful hemostasis rate is high, recurrent bleeding can occur, ranging from 10% to 50% according to the bleeding etiology. Therefore, how to reduce the rebleeding of GIB is an important clinical issue.

Methods: This is a randomized clinical trial. Patients with gastrointestinal bleeding for endoscopy screening and treatment at National Cheng Kung University Hospital were enrolled. The study will recruit 60 patients. After randomization, 30 patients will be classified into the intervention group and 30 into the control group. The participants will receive standard endoscopic hemostasis by either local injection of diluted epinephrine, heater probe coagulation, hemoclipping, or band ligation. After then, we will spray 2g of sucralfate powder and 1g of tranexamic acid through duodenoscopy precisely on the bleeding site in the intervention group. All enrolled patients will be monitored for rebleeding for 28 days after the first endoscopy.

DETAILED DESCRIPTION:
Gastrointestinal bleeding (GIB) is a common problem in the hospital. The annual rate of hospitalization for any type of GI hemorrhage is estimated to be 350 hospital admissions/100,000 population. GIB can be divided into upper GIB, small bowel bleeding, and lower GIB. Approximately 50% of admissions for GIB are for UGI bleeding (from the esophagus, stomach, and duodenum), 40% are for LGI bleeding (from the colon and anorectum), and 10% are for small intestine bleeding. Ulceration bleeding, variceal bleeding, angiodysplasia, Dieulafoy lesion, and tumor bleeding are common cause for UGIB, while diverticulosis, colitis, angioectasia, cancer bleeding, and polypectomy ulcer attribute to the LGIB. GI endoscopy can identify the bleeding site and permit therapeutic hemostasis in most patients with GI bleeding.

Endoscopic hemostasis includes epinephrine injection, hemoclipping, heat probe coagulation, and Argon plasma coagulation. Although the successful hemostasis rate is high, recurrent bleeding can occur, ranging from 10% to 50% according to the bleeding etiology. Therefore, how to reduce the rebleeding of GIB is an important clinical issue.

Tranexamic acid (TXA) is a well-known antifibrinolytic agent that inhibits fibrin degradation by binding to tissue plasminogen, thereby preventing blood clot lysis and reducing bleeding. A recent study evaluating the effect of topical tranexamic acid (TXA) powder on bleeding peptic ulcers demonstrated that the precise endoscopic administration of TXA powder can enhance the stop-bleeding effect.

Sucralfate, a complex of aluminum hydroxide and sucrose octa sulfate, can bind to the wound base. This protective barrier can prevent the wound from further environmental injury. Sucralfate has been widely used for wounds and ulcer treatment, e.g., skin wounds, oral ulcers, and peptic ulcers. With the protective effect of the papilla mucosa, sucralfate can cover the wound and has the potential to avoid further environmental damage. In combination with TXA powder in stabilizing the clotting, we expect the rebleeding event will reduce. Therefore, this study aimed to investigate whether the combination therapy of topical administration of TXA and sucralfate after standard endoscopic hemostasis can reduce the rebleeding event.

Furthermore, the adhesion time of the hemostasis powder at the bleeding site is also an unknown issue. High-dose barium enema use provides better clinical outcomes for initial hemostasis and long-term prevention of rebleeding than conservative therapy in LGIB. In combination of barium, the position of hemostasis powder can be identified by Xray.

Subjects and protocols Participants will be recruited from the volunteers with gastrointestinal bleeding at National Cheng Kung University Hospital. Eligible participants include patients aged ≥ 18 years who accept endoscopy for GIB, including hematemesis, Tarry stool, or bloody stool. Patient consent forms will be given and explained to all patients before the endoscopy. Exclusion criteria include patients with no need of endoscopic hemostasis, allergy to sucralfate, tranexamic acid, or barium, pregnancy, and patients with hollow organ perforation. After patient enrollment, we will randomize the patient into either the intervention group or control group by sealed envelope randomization method.

After the standard endoscopic hemostasis by either epinephrine injection, hemoclipping, heat coagulation, or band ligation, we will randomly assign the patients to either a control or an intervention group. After then, we will spray 2g of sucralfate powder, 1g of tranexamic acid powder, and 1g of barium through the endoscopy precisely on the bleeding site in the intervention group.

Blood tests As ward routine for bleeding patient, a blood sample is obtained to measure creatinine, albumin, total bilirubin, hemoglobin, platelet, prothrombin time (PT), and activated partial thromboplastin time (APTT). All lab data are checked by the central laboratory of the National Cheng Kung University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants include patients aged ≥ 18 years who accept endoscopy for GIB, including hematemesis, Tarry stool, or bloody stool

Exclusion Criteria:

* no need of endoscopic hemostasis
* allergy to sucralfate, tranexamic acid, or barium
* pregnancy
* patients with hollow organ perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
the recurrent rate of GI bleeding during the study period | 28 days
  Recurrent bleeding was defined as remarkable hematochezia or Tarry stool with endoscopic evidence of the same site bleeding.

SECONDARY OUTCOMES:
the rate of rebleeding requiring transarterial embolization or emergency surgery | 28 days
  rebleeding requiring transarterial embolization or emergency surgery
length of hospitalization | 28 days
  length of hospitalization
all-cause mortality rate | 28 days
  all-cause mortality
adverse events rate from powder spray | 28 days
  adverse events from powder spray, such as perforation or thrombotic events

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The IPD will be shared once the trial completed and study published

REFERENCES:
- [Background] Saydam SS, Molnar M, Vora P. The global epidemiology of upper and lower gastrointestinal bleeding in general population: A systematic review. World J Gastrointest Surg. 2023 Apr 27;15(4):723-739. doi: 10.4240/wjgs.v15.i4.723. PMID 37206079
- [Background] Chiang HC, Chen PJ, Yang EH, Hsieh MT, Shih IC, Cheng HC, Chang WL, Chen WY, Chiu HC, Kuo HY, Tsai WC, Lo YN, Yang KC, Chiang CM, Chen WC, Huang KK, Tseng HH, Chen CY, Lin XZ, Chuang CH. Precise application of topical tranexamic acid to enhance endoscopic hemostasis for peptic ulcer bleeding: a randomized controlled study (with video). Gastrointest Endosc. 2023 Nov;98(5):755-764. doi: 10.1016/j.gie.2023.06.013. Epub 2023 Jun 24. PMID 37356632
- [Background] Masuelli L, Tumino G, Turriziani M, Modesti A, Bei R. Topical use of sucralfate in epithelial wound healing: clinical evidences and molecular mechanisms of action. Recent Pat Inflamm Allergy Drug Discov. 2010 Jan;4(1):25-36. doi: 10.2174/187221310789895649. PMID 19832693
- [Background] Nagata N, Niikura R, Shimbo T, Ishizuka N, Yamano K, Mizuguchi K, Akiyama J, Yanase M, Mizokami M, Uemura N. High-dose barium impaction therapy for the recurrence of colonic diverticular bleeding: a randomized controlled trial. Ann Surg. 2015 Feb;261(2):269-75. doi: 10.1097/SLA.0000000000000658. PMID 25569028